CLINICAL TRIAL: NCT06603831
Title: Randomized, Prospective and Multicenter Clinical Study for the Clinical Evaluation and Cost-effectiveness Analysis of 3D Digital Surgery in Traumatology and Orthopedic Surgery
Brief Title: Clinical Evaluation and Cost-effectiveness Analysis of 3D Digital Surgery in Traumatology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital de Granollers (Other); Fundació Hospital d'Olot i Comarcal de la Garrotxa (Unknown); Hospital de la Santa creu i Sant Pau - Barcelona (Other); Consorci Hospitalari de Vic (Other); Corporació de Salut del Maresme i la Selva (Other)
Responsible Party: Principal Investigator, Ferran Fillat Gomà, Principal Investigator, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3DAdopt
Record Dates: First submitted 2024-07-22; First posted 2024-09-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Radius; Deformity; Hip Osteoarthritis; Hip Arthritis; Hip Arthropathy; Spine Injury; Radius; Anomaly; Vertebra; Degeneration; Vertebral Fracture; Hip Prosthesis Infection; Spinal Fusion; Spine Osteoarthritis; Spinal Deformity
MeSH Terms: conditions — Congenital Abnormalities; Osteoarthritis, Hip; Spinal Injuries; Spinal Fractures; Osteoarthritis, Spine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D digital surgery group (Experimental)
  Interventions: Procedure: patients treated using 3D technology and Patient-Specific Instrumentation
- 2D conventional surgery group (Active Comparator)
  Interventions: Procedure: Patients treated with conventional surgery, without using 3D technology

INTERVENTIONS:
Procedure: patients treated using 3D technology and Patient-Specific Instrumentation — 3D Digital surgery includes:
  * 3D Surgical Planning using biomedical engineering software; 3D visualization of the patients anatomy and surgical simulation.
  * Use of personalized surgical guides created through additive manufacturing.
  * Use of personalized implants created through additive manufacturing.
    3 surgical procedures are studied in this study; radius osteotomy, acetabular arthroplasty and spinal arthrodesis
  Arms: 3D digital surgery group
Procedure: Patients treated with conventional surgery, without using 3D technology — Conventional surgery includes:
  * 2D planning using TC and x-rays
  * Free-hand surgery
  * Use of generic, non-personalized implants
    3 surgical procedures are studied in this study; radius osteotomy, acetabular arthroplasty and spinal arthrodesis
  Arms: 2D conventional surgery group

SUMMARY:
Digital surgery, in combination with patient specific instrumentation (PSI) is being used more and more in traumatology due to its proven benefits and applications. Nowadays, medical case planning and an optimal preparation before surgery are still a challenge for surgeons. This lack of preparation is translated into longer surgical procedures, potential complications, unnecessary sterilization of materials and a high number of fluoroscopies. 2D techniques such as Magnetic Resonance Imaging (MRI), Computed Tomography (CT) and X-rays remain essential for medical planning, however, in many cases, a 3D visualization is needed to achieve better results, especially in complex cases.The use of personalized medical instruments such as surgical guides has proven to increase clinical accuracy, assuring a better correction of bone deformities, and allowing a more precise location of implants and screw positioning. Furthermore, the use of 3D-printed patient-specific prosthesis can lead to better clinical outcomes as they reduce the number of complications as well as they present a longer lifespan compared to conventional generic implants.Despite the potential of 3D technology in the medical field, there is still a lack of robust studies that compares clinical benefits between digital surgery and conventional 2D surgery, and its economic impact is still unknown. Thus, the investigators propose this randomized, prospective and multi-center clinical study to evaluate the use of 3D technology in traumatology. The aim of this project is to prove that digital surgery is a cost-effective methodology and therefore it should be adopted by the public health system as a gold standard procedure.

DETAILED DESCRIPTION:
3D technology is increasingly being used, especially in orthopaedic surgery and traumatology as it allows to define specific objects and to understand structures and system dynamics. From patient TC images and using a biomedical engineering software, an exact 3D virtual model of the anatomical region can be created, enabling visualization, planning and simulation of the entire surgery. Besides, this software allows to design custom-made surgical guides (that precisely define cutting zones and screw positioning) as well as personalized implants that perfectly fit the patient's anatomy. After that, Patient-Specific Instrumentation can be manufactured using 3D printers and biocompatible materials and they can be sterilized to be used in the operating room.

While personalized surgical guides increase surgical precision and surgeon satisfaction, personalized implants have shown to generate better clinical outcomes, both short and long term. Despite of the benefits that 3D technology can generate in the medical field, most surgeons still opt for conventional 2D planning techniques, free-hand surgeries and generic implants use. This results in a non-standardized and variable procedure that heavily depends on the surgeon´s experience and in many cases, the obtained results deviate from the initial goals. Scientific evidence shows that a lack of precision is strictly related to clinical complications. Poor alignment of the implants can cause damage to internal structures, increases chances of dislocations, fractures and osteolysis as well as reduces the prosthetic component lifespan. That translates into patient suffering from chronic pain, reduced functionality and an increased number of reinterventions.

Regardless of the potential and several applications of 3D technology, there´s still a lack of clinical evidence, and the economic impact is still unknown. This methodology is increasingly being used as a routine medical process in many institutions but still raises concerns regarding costs, specially when considering its use in the public health system. Although digital surgery has a wide variety of associated expenses such as hardware and software cost, equipment maintenance and 3D-specialised engineers, the cost of 3D technology has significantly decreased in the past few years and it can potentially generate economic benefits compared to the standard methodology due to the optimization of the surgical process; shorter surgeries, reduced number of unnecessary sterilized materials, reduced number of fluoroscopies during surgery and less medical complications and revisions.

Thus, a large-scale study is still needed to demonstrate: 1) clinical benefits that 3D technology can generate compared to conventional surgery and 2) thoroughly analyse its economic impact to determine if it's a cost-effective methodology. For this reason, a multi-centre, randomized and prospective study is proposed to evaluate digital surgery's clinical results and to perform a cost-effectiveness analysis in order to obtain enough scientific evidence to be able to escalate the use of 3D technology in all public health institutions.

This clinical trial is a pragmatic study that will evaluate the efficacy and effectiveness of 3D technology in 3 different surgical procedures; distal radius osteotomy, acetabular arthroplasty and spinal arthrodesis.

ELIGIBILITY:
Inclusion Criteria:

- Patients that requires one of the following surgical procedures / interventions: Radius osteotomy due to non-articular metaphyseal malunion Complex acetabular arthroplasty Thoracic-lumbar spine arthrodesis.

-Patients that can understand the clinical study and that are able to read, understand and sign the consent form

Exclusion Criteria:

* Patients that are not able to read, understand or sign the consent form.
* Patients that can't or have no support to complete the clinical trial.
* Patients with complex deformities or complications that would require mandatory personalized digital surgery treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of implants location, screw positioning and correction angles in regards the previous clinical planning and positioning reference standards. | CT will be performed before surgery and after 21 days of surgery. From this CT, positioning and correction measurements will be obtained in the lab and accuracy will be deduced.
  CT scan will be performed before and after surgery. Digital Planning will be performed in all cases to determine the right positioning of implants and screws (and deformity angle correction if needed) that the surgeon should achieve. Implant location and screw positioning from post-surgery CT will be measured and accuracy will be obtained by comparing the final positioning and correction with the previous planning and goals. Positioning and corrections measurements in post-surgery CT Scan will also be compared to positioning reference standards to determine the number of cases where the reference safe zone positioning and corrections have been achieved in both, digital and conventional surgery.

SECONDARY OUTCOMES:
Demographic | During patient recruitment
Pain of patient that undergoes any of the surgical procedures studied in this trial before and after surgery assessed by BPI-SF | This outcome will be measured before surgery, 21 days after surgery and 12 months after surgery
  Pain will be assessed by BPI-SF before and after surgery and results will be compared between digital and conventional surgery to determine if there are significant results in these clinical outcomes.
Quality of life of patients that undergoes any of the surgical procedures studied in this trial before and after surgery will be assessed by SF-36 questionnaire | This outcome will be measured before surgery, 21 days after surgery and 12 months after surgery
  Quality of life will be assessed by SF-36 before and after surgery and results will be compared between digital and conventional surgery to determine if there are significant results in these clinical outcomes.
Quality of life of patients that undergoes any of the surgical procedures studied in this trial before and after surgery will be assessed by EQ5D-5L questionnaire | This outcome will be measured before surgery, 21 days after surgery and 12 months after surgery
  Quality of life will be assessed by EQ5D-5L before and after surgery and results will be compared between digital and conventional surgery to determine if there are significant results in these clinical outcomes.
Functionality and pain for patients that undergoes radial osteotomy will be assessed by the specific PROM questionnaire PRWE | This outcome will be measured before surgery, 21 days after surgery and 12 months after surgery
  PRWE it's a patient reported outcome measures (PROMs) designed to measure wrist pain and disability in activities of daily living used for specific wrist problems
Functionality and pain for patients that undergoes hip arthroplasty will be assessed by the specific PROM questionnaire HOOS | This outcome will be measured before surgery, 21 days after surgery and 12 months after surgery
  HOOS it's a patient reported outcome measures (PROMs) designed to evaluate symptoms and limitations for patients with hip pain.
Functionality and pain for patients that undergoes spinal arthrodesis will be assessed by the specific PROM questionnaire Oswerty scale | This outcome will be measured before surgery, 21 days after surgery and 12 months after surgery
  Oswerty scale it's a patient reported outcome measure (PROMs) designed to evaluate pain and disability for patients that undergo arthrodesis and it's the gold standard of low back functional outcome tools.
Number of doctors and professionals that are present in the operating room | During surgery
  Outcome associated with surgery cost
surgical time. Length of time for the whole surgical intervention | During surgery
  Outcome associated with surgery cost
Post-operative time. Length of time for the whole post-operative procedure. | up to 1 day
  Outcome associated with surgery cost
number of surgical sets and sterilized material that has been used during surgery | During surgery
  Outcome associated with surgery cost
Complications that the patient can suffer during surgery | During surgery
  Any incidence that can happen to the patient during the whole intervention
Amount of fluoroscopies measured in fluoroscopy scan time that is used during surgery | During surgery
  measure the amount of fluoroscopies that the surgeon needed during the intervention.
number of medical follow-up visits or hospital resources | 1 year
  medical visits that the patient needs after surgery. this outcome is associated with cost.

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Fillat-Gomà, Principal Investigator — Corporacion PT
Locations (1):
- Hospital Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The plan is to create a data repository with all the outcomes obtained during this study for each patient.
  Study results will be also published in scientific reviews.
Supporting Information: SAP, CSR
Time Frame: Data will be available when the study is completed and will be shared for a minimum of 25 years

REFERENCES:
- [Background] Hoang D, Perrault D, Stevanovic M, Ghiassi A. Surgical applications of three-dimensional printing: a review of the current literature & how to get started. Ann Transl Med. 2016 Dec;4(23):456. doi: 10.21037/atm.2016.12.18. PMID 28090512
- [Background] Song Z, Dong W, Yang D, Yang J, Wu J, Wang Y, Gu Y. Application of 3D Visualization Technology in Complex Abdominal Wall Defects. Int J Gen Med. 2021 Jun 10;14:2449-2457. doi: 10.2147/IJGM.S310170. eCollection 2021. PMID 34140800
- [Background] Wang Y, Cao D, Chen SL, Li YM, Zheng YW, Ohkohchi N. Current trends in three-dimensional visualization and real-time navigation as well as robot-assisted technologies in hepatobiliary surgery. World J Gastrointest Surg. 2021 Sep 27;13(9):904-922. doi: 10.4240/wjgs.v13.i9.904. PMID 34621469
- [Background] Zoabi A, Redenski I, Oren D, Kasem A, Zigron A, Daoud S, Moskovich L, Kablan F, Srouji S. 3D Printing and Virtual Surgical Planning in Oral and Maxillofacial Surgery. J Clin Med. 2022 Apr 24;11(9):2385. doi: 10.3390/jcm11092385. PMID 35566511
- [Background] Lal H, Patralekh MK. 3D printing and its applications in orthopaedic trauma: A technological marvel. J Clin Orthop Trauma. 2018 Jul-Sep;9(3):260-268. doi: 10.1016/j.jcot.2018.07.022. Epub 2018 Aug 3. PMID 30202159
- [Background] Fillat-Goma F, Marcano-Fernandez FA, Coderch-Navarro S, Martinez-Carreres L, Berenguer A. 3D printing innovation: New insights into upper extremity surgery planning. Injury. 2021 Jul;52 Suppl 4:S117-S124. doi: 10.1016/j.injury.2021.01.048. Epub 2021 Feb 13. PMID 33632605
- [Background] Tallarico M, Scrascia R, Annucci M, Meloni SM, Lumbau AI, Koshovari A, Xhanari E, Martinolli M. Errors in Implant Positioning Due to Lack of Planning: A Clinical Case Report of New Prosthetic Materials and Solutions. Materials (Basel). 2020 Apr 16;13(8):1883. doi: 10.3390/ma13081883. PMID 32316361
- [Background] Myers CA, Laz PJ, Shelburne KB, Judd DL, Huff DN, Winters JD, Stevens-Lapsley JE, Rullkoetter PJ. The impact of hip implant alignment on muscle and joint loading during dynamic activities. Clin Biomech (Bristol). 2018 Mar;53:93-100. doi: 10.1016/j.clinbiomech.2018.02.010. Epub 2018 Feb 14. PMID 29482087
- [Background] Kim YH, Park JW, Kim JS, Park SD. The relationship between the survival of total knee arthroplasty and postoperative coronal, sagittal and rotational alignment of knee prosthesis. Int Orthop. 2014 Feb;38(2):379-85. doi: 10.1007/s00264-013-2097-9. Epub 2013 Sep 10. PMID 24173677
- [Background] Michielsen M, Van Haver A, Bertrand V, Vanhees M, Verstreken F. Corrective osteotomy of distal radius malunions using three-dimensional computer simulation and patient-specific guides to achieve anatomic reduction. Eur J Orthop Surg Traumatol. 2018 Dec;28(8):1531-1535. doi: 10.1007/s00590-018-2265-0. Epub 2018 Jun 20. PMID 29926244
- [Background] Coakley M, Hurt DE. 3D Printing in the Laboratory: Maximize Time and Funds with Customized and Open-Source Labware. J Lab Autom. 2016 Aug;21(4):489-95. doi: 10.1177/2211068216649578. Epub 2016 May 19. PMID 27197798
- [Background] Ballard DH, Mills P, Duszak R Jr, Weisman JA, Rybicki FJ, Woodard PK. Medical 3D Printing Cost-Savings in Orthopedic and Maxillofacial Surgery: Cost Analysis of Operating Room Time Saved with 3D Printed Anatomic Models and Surgical Guides. Acad Radiol. 2020 Aug;27(8):1103-1113. doi: 10.1016/j.acra.2019.08.011. Epub 2019 Sep 18. PMID 31542197
- [Background] Levesque JN, Shah A, Ekhtiari S, Yan JR, Thornley P, Williams DS. Three-dimensional printing in orthopaedic surgery: a scoping review. EFORT Open Rev. 2020 Aug 1;5(7):430-441. doi: 10.1302/2058-5241.5.190024. eCollection 2020 Jul. PMID 32818070
- [Background] von Campe A, Nagy L, Arbab D, Dumont CE. Corrective osteotomies in malunions of the distal radius: do we get what we planned? Clin Orthop Relat Res. 2006 Sep;450:179-85. doi: 10.1097/01.blo.0000223994.79894.17. PMID 16721354
- [Background] Delbruck H, Weber DC, Eschweiler J, Hildebrand F. 3D accuracy and clinical outcomes of corrective osteotomies with patient-specific instruments in complex upper extremity deformities: an approach for investigation and correlation. Eur J Med Res. 2022 Oct 8;27(1):197. doi: 10.1186/s40001-022-00830-9. PMID 36209123
- [Background] Tack P, Victor J, Gemmel P, Annemans L. Do custom 3D-printed revision acetabular implants provide enough value to justify the additional costs? The health-economic comparison of a new porous 3D-printed hip implant for revision arthroplasty of Paprosky type 3B acetabular defects and its closest alternative. Orthop Traumatol Surg Res. 2021 Feb;107(1):102600. doi: 10.1016/j.otsr.2020.03.012. Epub 2020 May 11. PMID 32409268
- [Background] Lewinnek GE, Lewis JL, Tarr R, Compere CL, Zimmerman JR. Dislocations after total hip-replacement arthroplasties. J Bone Joint Surg Am. 1978 Mar;60(2):217-20. PMID 641088
- [Background] Buller L, Smith T, Bryan J, Klika A, Barsoum W, Iannotti JP. The use of patient-specific instrumentation improves the accuracy of acetabular component placement. J Arthroplasty. 2013 Apr;28(4):631-6. doi: 10.1016/j.arth.2012.12.001. PMID 23498350
- [Background] Gertzbein SD, Robbins SE. Accuracy of pedicular screw placement in vivo. Spine (Phila Pa 1976). 1990 Jan;15(1):11-4. doi: 10.1097/00007632-199001000-00004. PMID 2326693
- [Background] Zhang XN, Zhou LJ, Su QJ, Guan L, Li DY, Pei BQ, Pan AX, Yang HH, Ding HT, Liu YZ, Hai Y. Accuracy of cortical bone trajectory screw fixation guided by spinous process clamp guide in lumbosacral vertebrae: A cadaver study. Int J Med Robot. 2023 Apr;19(2):e2484. doi: 10.1002/rcs.2484. Epub 2022 Dec 16. PMID 36413096
- [Background] Maruo K, Arizumi F, Kusuyama K, Kishima K, Tachibana T. Accuracy and safety of cortical bone trajectory screw placement by an inexperienced surgeon using 3D patient-specific guides for transforaminal lumbar interbody fusion. J Clin Neurosci. 2020 Aug;78:147-152. doi: 10.1016/j.jocn.2020.04.090. Epub 2020 Apr 27. PMID 32354646
- [Background] Phan K, Sgro A, Maharaj MM, D'Urso P, Mobbs RJ. Application of a 3D custom printed patient specific spinal implant for C1/2 arthrodesis. J Spine Surg. 2016 Dec;2(4):314-318. doi: 10.21037/jss.2016.12.06. PMID 28097249